CLINICAL TRIAL: NCT05565209
Title: Left Atrial Appendage Closure Registry of Henri Mondor Hospital
Acronym: FLAAC3
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220614
Record Dates: First submitted 2022-09-15; First posted 2022-10-04 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation, Left atrial appendage closure, stroke, anticoagulation, bleeding
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SA brief descriptive name used to refer to the intervention(s) studied — Details that can be made public about the intervention

SUMMARY:
Intro: Patients with atrial fibrillation are at significant risk of thrombus formation in the left atrial appendage, which can lead to strokes or systemic embolisms. This risk justifies first-line prescribing of long-term oral anticoagulant therapy in these patients. Percutaneous left atrial appendage closure, is an interventional cardiology technique for patients at high risk of stroke related to atrial fibrillation in whom long term anticoagulation therapy cannot be conducted. This procedure involves implantation of an occlusion device into the left atrial appendage to close it and prevent migration of thrombotic material that could otherwise cause distant embolism. Closure of the left atrial appendage avoids long-term prescription of anticoagulants while protecting patients against the risk of systemic embolism and stroke.

Hypothesis/Objective: the main objective of this study is to assess the long term efficacy of left atrial closure, 5 years after the procedure Method: 150 patients will be included prospectively. We will also include restropectively100 other patients, previously treated by left atrial appendage closure at Henri Mondor hospital. Demographic, clinical, echocardiographic, and computed tomography data will be obtained by physical examination or medical records.

Conclusion: this study will allow to assess the long term efficacy of left atrial closure in atrial fibrillation patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patient for whom an indication has been made for implantation of a device for the closure of the left atrial appendage without restriction of indication and regardless of the outcome of the procedure (implantation success or not)

Exclusion Criteria:

* Refusal of the patient to participate in this study
* Minor patient
* Patient not affiliated to the French social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A description of the population from which the groups or cohorts will be selected
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-09-24 (Actual); Primary Completion 2026-09-14 (Estimated); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
Frequency of thrombo-embolic events | 60months of follow-up after the procedure
  The primary efficacy endpoint is the frequency of a combined endpoint including ischemic strokes and systemic embolisms after left atrial appendage closure. This frequency will be expressed as the percentage of patients who presented at least one of these events. Only the first event occurring in each patient will be taken into account, in the case where the same patient would present several events.

SECONDARY OUTCOMES:
Efficacy of the procedure | One hour after the end of the procedure
  : At the end of the procedure, the efficiency of the procedure will be described by the percentage of success of the procedure. The successful procedure is defined by a successful implantation of the device in the left atrial appendage without presaging its occlusive character.
  One hour after the end of the procedure
Occlusion of the left atrial appendage | 3 months
  The percentage of left atrial appendage occlusion is defined as the percentage of patients where left atrial appendage is efficiently closed at by transesophageal echography and / or CT scan Time Frame: 3 months
residual peri-device leak | 3 months
  The percentage a patients with 3 months residual peri-device leak will be determined at transesophageal echography and / or CT scan
Percentage of ischemic stroke | 1 and 5 years after the procedure
  Percentage of patients with at least one ischemic stroke during the study
Percentage of transient ischemic attack (TIA) | 1 and 5 years after the procedure
  Percentage of patients presenting at least one systemic embolism during the study
Percentage of systemic embolism | 1 and 5 years after the procedure
  Percentage of patients presenting at least one systemic embolism during the study
Cardiovascular or unexplained death | 1 and 5 years after the procedure
  Percentage of patients who had a cardiovascular or unexplained death during the study
All-cause mortality | 1 and 5 years after the procedure
  percentage of all cause deaths
Comparison of the rate of thromboembolic events to expected values | 1 and 5 years after the procedure
  the observed rate of thromboembolic event will be compared to the expected value, according the individual patients CHA2DS2-VASc scores
Rate of complications related or potentially related to the device or the implantation procedure | periprocedural period (defined as the time from the day of the procedure to day 7 or discharge, whichever comes last)
  : Rate of complications related or potentially related to the device or the implantation procedure
Percentage of pericardial effusion | Periprocedural period (defined as the time from the day of the procedure to day 7 or discharge, whichever comes last)
  Percentage of patients who presented a pericardial effusion objectified by trans-thoracic ultrasound
Percentage of pericardial effusion | 3 months
  Percentage of patients who presented a pericardial effusion objectified by trans-thoracic ultrasound
Percentage of migration of the device | periprocedural period (defined as the time from the day of the procedure to day 7 or discharge, whichever comes last)
  Percentage of patients who presented a migration of the device, objectified by echocardiography and / or CT scan
Percentage of migration of the device | 3 months; 1 year; 5 years
  : Percentage of patients who presented a migration of the device, objectified by the echocardiography and / or CT scan
Percentage of device thrombosis | 3 months; 1 year; 5 year
  Percentage of patients who presented a thrombosis on the device, objectified by transesophageal echography and / or CT scan
Bleeding (all cause) | 1 year; 5 year
  Percentage of patients who presented a bleeding
Bleedings not-related to the procedure or the device | 1 year; 5 year
  Percentage of patients who presented a bleeding not-related to the procedure or the device
Criteria for Evaluating Associated Antithrombotic Treatments | : Discharge, 3, 6, 12 months after the procedure, 1 and 5 years after the procedure
  The antithrombotic treatments will be collected at different follow-up times.
  The type and duration of anti-thrombotic treatments will be documented using the combined criteria:
  * Percentage of patients on injectable or oral anticoagulants and antiplatelet agents at different follow-up times
  * Percentage of patients on injectable or oral anticoagulants at different follow-up times
  * The percentage of patients on platelet antiaggregants in single or dual therapy at different follow-up times
Description of the population | At inclusion
  Demographic and clinical characteristics of the patients will be collected and described, such as: age, sex, medical and surgical history, cardiovascular pharmacological treatments, comorbidities, indication of left atrial closure, HAS-BLED and CHA2DS2-VASc scores, anatomical features of the left atrial appendage at inclusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION